CLINICAL TRIAL: NCT04410198
Title: A Phase 3b Multicenter, Open-Label Single Arm Study of Roxadustat: Either as Conversion From a Continuous Erythropoietin Receptor Activator (CERA), or as Initial Anemia Treatment in Hemodialysis (HD) Patients - DENALI Study
Brief Title: Study of Roxadustat Conversion in Participants Receiving Stable Erythropoiesis-Stimulating Agent (ESA) or as Initial Anemia Treatment in Chronic Dialysis Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-097
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Anemia Associated With End Stage Renal Disease (ESRD)
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Roxadustat (Experimental): Participants will receive roxadustat as an oral tablet, 3 times per week (TIW) for up to a maximum of 24 weeks. If a participant requires roxadustat <60 milligrams (mg)/week to maintain Hb levels, the dose frequency will be reduced in a stepwise manner, for example, to BIW, and then QW. For participants converted from CERA, the initial roxadustat dose will be based on the average prescribed CERA dose in the last 8 weeks prior to conversion. For participants with <6 weeks of prior CERA use, the initial roxadustat dose will be based on a 2-tiered, weight-based dosing scheme. Dose adjustment evaluations will be made every 4 weeks and doses will be titrated based on Hb level and rate of Hb change. The prescribed dose will not exceed the maximum allowable dose of 3.0 mg/kilogram (kg)/dose or 400 mg per dose, whichever is lower.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be administered per dose and schedule specified in the arm description.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of Roxadustat dosing regimens among chronic dialysis participants converted from ESA therapy or who are ESA-naïve.

ELIGIBILITY:
Key Inclusion Criteria:

* Receiving chronic dialysis for end stage renal disease (ESRD)
* Vascular access must be a functioning native arteriovenous fistula or graft with adequate flow in the opinion of the investigator, or permanent tunneled catheter
* Screening hemoglobin criteria (based on central lab value; measured within 10 days prior to initiating Roxadustat treatment: Participants converting from CERA: screening heamoglobin was between 9.0 to 12.0 g/dL; Participants initiating anemia treatment: <10.0 g/dL
* Ferritin ≥ 50 nanograms (ng)/milliliter (mL), Transferrin saturation (TSAT) ≥ 10% at screening
* Participant's alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are ≤3 x upper limit of normal (ULN), and total bilirubin (TBL) is ≤1.5 x ULN at screening and prior to initiating roxadustat treatment.
* Body weight between 45.0 to 160.0 kg

Key Exclusion Criteria:

* Red blood cell (RBC) transfusion within 4 weeks prior to enrollment
* Known history of myelodysplastic syndrome or multiple myeloma
* Known hereditary hematologic disease or other known causes for anemia other than chronic kidney disease (CKD)
* Known chronic inflammatory disease that is determined by the investigator to be the primary cause of anemia
* Active or chronic gastrointestinal bleeding
* Treated with iron-chelating agents within 4 weeks prior to enrollment
* History of New York Heart Association (NYHA) Class III or IV congestive heart failure
* History of myocardial infarction (MI), acute coronary syndrome, stroke, seizure, or a thrombotic/thromboembolic event (excluding vascular dialysis access stenosis/thrombosis) within 12 weeks prior to enrollment
* Uncontrolled hypertension, in the opinion of the Investigator
* Diagnosis or suspicion of renal cell carcinoma as shown on renal imaging performed within 24 weeks prior to enrollment
* History of malignancy, except for cancers determined to be cured or in remission for ≥2 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Eisner, Study Chair — Kyntra Bio
Locations (9):
- United States (9):
  - Investigational Site, Englewood, Colorado
  - Investigational Site, Caldwell, Idaho
  - Investigational Site, Baton Rouge, Louisiana
  - Investigational Site, Kalamazoo, Michigan
  - Investigational Site, Tupelo, Mississippi
  - Investigational Site, Saint Ann, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Sugar Land, Texas
  - Investigational Site, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Roxadustat: Participants received roxadustat as an oral tablet, 3 times per week (TIW) for up to a maximum of 24 weeks. If a participant required roxadustat <60 milligrams (mg)/week to maintain hemoglobin (Hb) levels, the dose frequency was reduced in a stepwise manner, for example, to twice weekly (BIW), and then once weekly (QW). For participants converted from continuous erythropoietin receptor activator (CERA), the initial roxadustat dose was based on the average prescribed CERA dose in the last 8 weeks prior to conversion. For participants with <6 weeks of prior CERA use, the initial roxadustat dose was based on a 2-tiered, weight-based dosing scheme. Dose adjustment evaluations were made every 4 weeks and doses were titrated based on Hb level and rate of Hb change. The prescribed dose did not exceed the maximum allowable dose of 3.0 mg/kilogram (kg)/dose or 400 mg per dose, whichever was lower.
Period: Overall Study
Arm/Group | Roxadustat
Started | 203
Received at Least 1 Dose of Study Drug | 203
Full Analysis Set (All enrolled participants who provided baseline Hb data and data for at least 1 postbaseline Hb time point.) | 201
Completed | 166
Not Completed | 37
Not completed — Death | 10
Not completed — Withdrawal by Subject | 7
Not completed — Transferred/Relocation | 4
Not completed — Kidney Transplant | 9
Not completed — Adverse Event | 4
Not completed — Physician Decision | 2
Not completed — Other than specified | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Roxadustat: Participants received roxadustat as an oral tablet, TIW for up to a maximum of 24 weeks. If a participant required roxadustat <60 mg/week to maintain Hb levels, the dose frequency was reduced in a stepwise manner, for example, to BIW, and then QW. For participants converted from CERA, the initial roxadustat dose was based on the average prescribed CERA dose in the last 8 weeks prior to conversion. For participants with <6 weeks of prior CERA use, the initial roxadustat dose was based on a 2-tiered, weight-based dosing scheme. Dose adjustment evaluations were made every 4 weeks and doses were titrated based on Hb level and rate of Hb change. The prescribed dose did not exceed the maximum allowable dose of 3.0 mg/kg/dose or 400 mg per dose, whichever was lower.
Arm/Group | Roxadustat
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 168
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 84
  Race: American Indian or Alaska Native | 3
  Race: Asian | 4
  Race: Native Hawaiian or Other Pacific Islander | 3
  Race: White | 105
  Race: Other | 4
Baseline Hb [Mean (Standard Deviation); unit: grams (g)/deciliter (dL)] — Population: Here, Number analyzed = Participants evaluable for this baseline measure.
  grams (g)/deciliter (dL)
    number analyzed (Participants) | 202
    (all) | 10.402 (0.8159)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Mean Hb Value ≥10 g/dL
Description: Percentage of participants with mean Hb value ≥10 g/dL, averaged from Week 16 through Week 24 has been reported. 95% confidence interval (CI) was calculated based on the normal approximation to the binomial distribution.
Time Frame: Week 16 through Week 24
Population: The full analysis set included all enrolled participants who provided baseline Hb data and data for at least 1 postbaseline Hb time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 201
percentage of participants | 84.7 [79.1 to 90.2]

2. Primary Outcome: Mean Hb Change From Baseline to Average Hb From Weeks 16-24
Description: Baseline Hb was defined as the mean of available central laboratory Hb values prior to first dose of study medication including the predose Hb value collected on Day 1. Missing data was imputed using Monte Carlo Markov Chain (MCMC) imputation model.
Time Frame: Baseline, Weeks 16-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat
Number analyzed (Participants) | 201
g/dL | 0.46 (1.007)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days post last dose of roxadustat (Week 28)
Description: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Arm/Group | Roxadustat
All-Cause Mortality (participants affected / at risk) | 10/203
Serious Adverse Events (participants affected / at risk) | 52/203
Other Adverse Events (participants affected / at risk) | 34/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=203)
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 4
Cardiac arrest (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Vitritis (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 3
Death (General disorders) | 2
Catheter site haemorrhage (General disorders) | 1
Hypothermia (General disorders) | 1
Medical device site haemorrhage (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pain (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
COVID-19 (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 4
Arteriovenous graft site infection (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Coronavirus infection (Infections and infestations) | 1
Endophthalmitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 1
Vascular access steal syndrome (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 2
Brain injury (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Post cardiac arrest syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Spinal cord infarction (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Device malfunction (Product Issues) | 1
Bipolar disorder (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Hypertensive urgency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=203)
Diarrhoea (Gastrointestinal disorders) | 15
COVID-19 (Infections and infestations) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04410198/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT04410198/SAP_001.pdf